CLINICAL TRIAL: NCT00535483
Title: An Open, Mono-centre Pilot Study to Investigate a Novel Technique to Establish Glycaemic Control for Critically Ill Patients, Tested in Type 1 Diabetic Subjects for a Period of 30 Hours.
Brief Title: Closed Loop Insulin Therapy in Type 1 Diabetics Based on Blood Microdialysis, Online Sensors and an eMPC Algorithm
Status: Completed | Type: Observational
Sponsor: Medical University of Graz (Other)
Other Study IDs: ABS3
Record Dates: First submitted 2007-09-24; First posted 2007-09-26 (Estimated); Last update posted 2014-04-04 (Estimated); Status verified 2014-04

CONDITIONS: Type 1 Diabetes
Keywords: blood microdialysis; glucose monitoring; glucose control; automated blood sampling; online-sensor; algorithm; type 1 diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The EU funded project CLINICIP (Closed Loop Insulin Infusion for Critically Ill Patients) aims to develop a low-risk monitoring and control device which allows maintaining metabolic control in intensive care units. A system will be developed comprising three subsystems: a body interface for the delivery of biofluids, biosensors for the determination of glucose concentration in these biofluids and an adaptive control algorithm that generates advice and thus represents a decision support system with respect to insulin infusion rate to establish glycaemic control in critically ill patients. Within a closed loop system, intensified insulin treatment will make use of the calculations leading to external regulation of glucose.

It is the aim of this study to evaluate the feasibility to establish glycaemic control in type 1 diabetic subjects over a period of 30 hours by manually combining these three - previously tested - subsystems (ABS System, extracorporeal online glucose sensor and a laptop-based computer algorithm).

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent obtained before any trial-related activities
* Age of analysable subjects in the range from 18 to 65 years
* Type 1 diabetes (Treatment with multiple daily injection for more than 12 months)

Exclusion Criteria:

* Severe acute and/or chronic diseases
* Mental incapacity, unwillingness or language barriers precluding adequate understanding or co-operation
* Taking of any vasoactive substances or anticoagulation medication.
* Diseases of the skin which could interfere with application of the catheters.
* Pregnancy or breastfeeding
* Bleeding disorder
* Known heparin allergy or heparin intolerance

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2007-08; Study Completion 2007-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas R Pieber, MD, Principal Investigator — Medical University Graz, Graz, Austria
Locations (1):
- Medical University Graz - Clinical Research Center, Graz, Styria, Austria

REFERENCES:
- See also: http://www.joanneum.at/health — http://www.joanneum.at/health